CLINICAL TRIAL: NCT05727241
Title: The Effect of Three-dimensional Umbilical Cord Coiling Index on Obstetrical and Neonatal Outcomes: a Prospective Study
Brief Title: Three-dimensional Umbilical Cord Coiling Index
Status: Not yet recruiting | Type: Observational
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, Dr Raneen Abu Shqara, Doctor, Western Galilee Hospital-Nahariya
Other Study IDs: 0080-22-NHR
Record Dates: First submitted 2023-02-04; First posted 2023-02-14 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Umbilical Cord Issue; Intrauterine Growth Restriction; Fetal Distress
Keywords: Coiling index; Neonatal outcome; Intrauterine Growth Restriction; Antepartum screening
MeSH Terms: conditions — Fetal Growth Retardation; Fetal Distress | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The study cohort (total sample): All women will undergo ultrasound examination for three-dimensional umbilical cord index.
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — The intervention is ultrasound examination with three dimensional umbilical cord index, two-dimensional umbilical cord index, and doppler examination of the umbilical cord artery.

SUMMARY:
Previous studies have shown that abnormal coiling of the umbilical cord is associated with adverse perinatal outcome. For example, an umbilical cord that is non-coiled increases the chance of fetal morbidity and mortality, moreover, they have shown that the lack of the usual coiled umbilical cord configuration may result in an umbilical cord that is structurally less able to withstand external mechanical stress, on the other hand, studies from recent years show that hypercoiling - excessive coiling of the umbilical cord is associated with poor obstetric outcomes, such as fetal distress at birth, meconium staining, fetal acidosis, premature birth, intrauterine growth disorder and even fetal death.

The studies carried out on the calculation of UCI include performing these measurements in two dimensions, including Doppler activation, but no studies were carried out in which three dimensions were used. The purpose of the study is to measure UCI using a 3D method in a random sample of 250 patients beyond 24 week of gestation, and to compare pregnancies with hypercoiling, hypocoiling or with a normal number of coils in terms of birth outcomes.

DETAILED DESCRIPTION:
The umbilical cord connects the growing fetus to the placenta and contains 3 blood vessels, 2 arteries and a vein. The umbilical cord is protected by a layer of Wharton jelly and is characterized by being coiled. This coiling provides the umbilical cord with strength and flexibility simultaneously, and as a result lowers the risk of complications such as torsion of the umbilical cord.

The reason for the formation of this coiling is unknown, but there are many hypotheses such as mobility and rotation of the fetus around the axis of the umbilical cord, a different growth pattern of the blood vessels in the umbilical cord and a special arrangement of the muscles in the walls of the arteries of the umbilical cord.

Umbilical cord index (UCI) is the distance between one coil of the umbilical cord. it is calculated from the inner edge of the wall of an umbilical cord artery or vein to the outer edge of the same vessel in the next coil, the direction is from the edge of the placenta to the fetus. The final value is the average of three readings in three different segments of the umbilical cord.

Previous studies have shown that abnormal coiling of the umbilical cord is associated with adverse perinatal outcome. For example, an umbilical cord that is non-coiled increases the chance of fetal morbidity and mortality, moreover, they have shown that the lack of the usual coiled umbilical cord configuration may result in an umbilical cord that is structurally less able to withstand external mechanical stress, on the other hand, studies from recent years show that hypercoiling - excessive coiling of the umbilical cord is associated with poor obstetric outcomes, such as fetal distress at birth, meconium staining, fetal acidosis, premature birth, intrauterine growth disorder and even fetal death.

The studies carried out on the calculation of UCI include performing these measurements in two dimensions, including Doppler activation, but no studies were carried out in which three dimensions were used. The purpose of the study is to measure UCI using a 3D method in a random sample of 250 patients beyond 24 week of gestation, and to compare pregnancies with hypercoiling, hypocoiling or with a normal number of coils in terms of birth outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Pregnancy week > or = 24.0

Exclusion Criteria:

* Twin pregnancy
* Pregnancy week<24
* Single umbilical cord
* Insufficient prenatal care
* Abnormal anatomical fetal findings, abnormal results of aneuploidy screening
* Premature rupture of membranes
* Polyhydramnios or Oligohydramnios at the time of recruitment.
* Intrauterine growth restriction at the time of recruitment

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The study is obstetrical
Study Population: This study will include low-risk singleton pregnancies, above 24 weeks of pregnancy, women with normal anatomical scan results and normal aneuploidy screening results. Women who have polyhydramnios, Oligohydramnios or intrauterine growth restriction at the time of recruitment will be ruled out.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Intrauterine growth restriction | 1 year
  The correlation between three-dimensional umbilical cord index and the rate of intrauterine growth restriction

SECONDARY OUTCOMES:
Two-dimensional umbilical cord index | 1 year
  The correlation between three-dimensional umbilical cord index and the two-dimensional umbilical cord index
Doppler index of the umbilical cord | 1 year
  The correlation between three-dimensional umbilical cord index and the doppler index of the umbilical cord
fetal distress during delivery | 2 years
  The correlation between three-dimensional umbilical cord index and the rate of fetal distress during delivery
Meconium staining | 2 years
  The correlation between three-dimensional umbilical cord index and meconium staining at delivery
Delivery mode | 2 years
  The correlation between three-dimensional umbilical cord index and the delivery mode
Cord pH | 2 years
  The correlation between three-dimensional umbilical cord index and Cord pH
APGAR score | 2 years
  The correlation between three-dimensional umbilical cord index and APGAR score
Newborn intensive care unit admission | 2 years
  The correlation between three-dimensional umbilical cord index and admission to NICU

CONTACTS AND LOCATIONS:
Overall Officials: Marwan Odeh, MD, Principal Investigator — Galilee Medical Center
Locations (1):
- Galilee Medical Center, Nahariya, Northern District, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chitra T, Sushanth YS, Raghavan S. Umbilical coiling index as a marker of perinatal outcome: an analytical study. Obstet Gynecol Int. 2012;2012:213689. doi: 10.1155/2012/213689. Epub 2012 Feb 14. PMID 22496697
- [Background] Ma'ayeh M, McClennen E, Chamchad D, Geary M, Brest N, Gerson A. Hypercoiling of the umbilical cord in uncomplicated singleton pregnancies. J Perinat Med. 2018 Aug 28;46(6):593-598. doi: 10.1515/jpm-2017-0034. PMID 28672757
- [Background] Strong TH Jr, Elliott JP, Radin TG. Non-coiled umbilical blood vessels: a new marker for the fetus at risk. Obstet Gynecol. 1993 Mar;81(3):409-11. PMID 8437796
- [Background] Degani S, Lewinsky RM, Berger H, Spiegel D. Sonographic estimation of umbilical coiling index and correlation with Doppler flow characteristics. Obstet Gynecol. 1995 Dec;86(6):990-3. doi: 10.1016/0029-7844(95)00307-d. PMID 7501354
- [Background] Sharma B, Bhardwaj N, Gupta S, Gupta PK, Verma A, Malviya K. Association of umbilical coiling index by colour Doppler ultrasonography at 18-22 weeks of gestation and perinatal outcome. J Obstet Gynaecol India. 2012 Dec;62(6):650-4. doi: 10.1007/s13224-012-0230-0. Epub 2012 Aug 17. PMID 24293842
- [Background] Rana J, Ebert GA, Kappy KA. Adverse perinatal outcome in patients with an abnormal umbilical coiling index. Obstet Gynecol. 1995 Apr;85(4):573-7. doi: 10.1016/0029-7844(94)00435-G. PMID 7898836
- [Background] Machin GA, Ackerman J, Gilbert-Barness E. Abnormal umbilical cord coiling is associated with adverse perinatal outcomes. Pediatr Dev Pathol. 2000 Sep-Oct;3(5):462-71. doi: 10.1007/s100240010103. PMID 10890931
- [Background] de Laat MW, Franx A, van Alderen ED, Nikkels PG, Visser GH. The umbilical coiling index, a review of the literature. J Matern Fetal Neonatal Med. 2005 Feb;17(2):93-100. doi: 10.1080/14767050400028899. PMID 16076615